CLINICAL TRIAL: NCT02905929
Title: Randomized Control Trial to Reduce Sitting Time in Postmenopausal Latina Women at Increased Risk for Heart Disease
Brief Title: Trial to Reduce Sitting Time in Postmenopausal Latina Women at Increased Risk for Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: South Bay Latino Research Center (Unknown); San Ysidro Health Center (Other); San Diego State University (Other)
Responsible Party: Principal Investigator, Matthew Allison, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 160682
Record Dates: First submitted 2016-09-09; First posted 2016-09-19 (Estimated); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Sedentary Lifestyle
Keywords: sedentary behavior; standing; sitting; inclinometer
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitting Less group (Experimental): The 'reduce sitting' intervention group will receive three in-person health coaching sessions followed by five counseling phone calls. Participants will wear a thigh worn inclinometer for the first 3 weeks of the intervention, and at the mid-point of the intervention. At each in-person health coaching session participants will receive feedback from the ActivPAL showing periods throughout the day where participants have been sitting. In addition to the three initial in-person counseling sessions using the ActivPAL feedback, participants will receive phone calls from the health educator biweekly to help overcome barriers, to work on self-monitoring and planning skills, and to prepare relapse prevention. Tools to help prompt standing, including a standing desk, will also be provided.
  Interventions: Device: ActivPAL inclinometer; Behavioral: Phone counseling call: Breaking up sitting time; Behavioral: In-person counseling: Breaking up sitting time; Other: Tools to prompt standing
- Attention Control (Active Comparator): Participants in the attention control condition will receive a healthy aging educational intervention developed and tested by the investigators in previous studies. This group will receive one in-person coaching session followed by seven phone coaching sessions.
  Interventions: Behavioral: Phone counseling call: Healthy living; Behavioral: In-person counseling: Healthy living

INTERVENTIONS:
Device: ActivPAL inclinometer — Participants will wear a thigh-worn inclinometer for the first 3 weeks of the intervention, and at the mid-point of the intervention. The device will monitor their sitting and standing time.
  Arms: Sitting Less group
Behavioral: Phone counseling call: Breaking up sitting time — Participants will receive 5 counseling phone calls to check-in on goal setting, strategies, and tools.
  Arms: Sitting Less group
Behavioral: In-person counseling: Breaking up sitting time — Participants will receive 3 in-person health education sessions. At these sessions participants will receive feedback from the ActivPAL showing periods throughout the day where participants have been sitting. Participants will also develop action plans, check-in on goal setting, and use of tools at these sessions.
  Arms: Sitting Less group
Behavioral: Phone counseling call: Healthy living — Participants will receive a healthy living educational intervention over the phone, developed and tested by the investigators in previous studies. Participants will not receive any information on diet, physical activity or sedentary behavior that may affect the outcomes.
  Arms: Attention Control
Other: Tools to prompt standing — Investigators will provide standing desks to participants who spend time sitting at a computer. Additional tools to help prompt standing are mechanical and electronic timers set to interrupt long periods of sitting and cues in the environment such as standing during commercial breaks and phone calls.
  Arms: Sitting Less group
Behavioral: In-person counseling: Healthy living — Control subjects will receive one in-person counseling session about healthy living. Participants will not receive any information on diet, physical activity or sedentary behavior that may affect the outcomes.
  Arms: Attention Control

SUMMARY:
Project 2 of the University of California, San Diego (UCSD) American Heart Association (AHA) Women's Health Program will assess 3-month changes in sitting time, standing time, physical activity and blood pressure in a randomized control trial (RCT). This 2-arm RCT will occur in the community with post menopausal Latina women (N=250) who spend at least 8 hrs/day sitting and have increased risk for cardiovascular disease through high BMI and other cardiometabolic risk factors. Women will be identified through the San Ysidro Health Center and assessed at the South Bay Latino Research Center.

DETAILED DESCRIPTION:
Project 2 will address the following aims:

1. Investigate the 3 month effect of the intervention to impact the primary behavioral outcomes of sitting, standing and stepping time assessed objectively by a thigh worn inclinometer (ActivPAL) in Latinas at risk for heart disease.
2. Investigate the 3 month effect of the intervention to impact the secondary health outcomes of blood pressure, depressive symptoms, and anthropometrics.
3. Explore the psychosocial & environmental mediators & moderators of changes in sitting time.

ELIGIBILITY:
Inclusion criteria for RCT (n=250):

1. Postmenopausal woman, no menstruation for at least 1 year, 55+ years of age.
2. Self-identify as Hispanic ethnicity, able to read and write in English or Spanish,
3. Ambulatory, medically stable, able to give informed consent, and safely complete the protocols.
4. Body Mass Index range of 25.0-45.0kg/m2.
5. Sedentary: Average >8 hours sitting/day, as measured by ActivPAL on 4+ days per week
6. Phone access (to receive counseling)

Prisoners will not be used for this study.

Exclusion criteria applicable only to the RCT intervention trial participants include:

1. Unable to complete the Short Physical Performance Battery.
2. Mental states that would preclude complete understanding of the protocol and compliance.
3. Active cancer or another serious chronic illness that may be associated with weight change
4. Body Mass Index <25.0 or >45.0kg/m2.
5. Use of insulin medications.
6. ≤ 8hr average daily sitting time, as measured by ActivPAL.
7. Participating in another clinical trial related to study outcomes (as determined by the PI).
8. Unable to wear devices

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 254 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Sitting, standing and stepping time | 3 months
  Change in daily time spent sitting, standing and stepping during waking hours as measured objectively by the ActivPAL

SECONDARY OUTCOMES:
Blood pressure | 3 months
  Change in blood pressure
Depressive symptoms | 3 months
  Change in depressive symptoms, measured with Center for Epidemiologic Studies Depression (CESD) short form. Scores greater than 10 indicate probable depressive symptoms.
Improvement in Quality of Life | 3 months
  Change in quality of life, measured with the EURO-QOL 5-D, a brief 5 item standard scale that has demonstrated validity in populations with diabetes and cardiovascular diseases.
Anthropometrics | 3 months
  Change in body mass index (BMI)
Psychosocial and environmental mediators: benefits and barriers | 3 months
  Investigators will use measures adapted for our pilot that include benefits and barriers to sitting less.
Psychosocial and environmental mediators: self-efficacy | 3 months
  Investigators will use measures adapted for our pilot including self-efficacy to sit less.
Psychosocial and environmental mediators: social support | 3 months
  Investigators will use measures adapted for our pilot including social support surrounding sitting less.
Psychosocial and environmental mediators: home environment support | 3 months
  Investigators will use measures adapted for our pilot including home environment support surrounding sitting less.
Psychosocial and environmental mediators: habit formation | 3 months
  Assessed using the Self-Report Habit Index
Demographic moderators: age | 3 months
  Self-reported items on the baseline survey. Some of these demographic variables will also be considered covariates in analyses.
Demographic moderators: sex | 3 months
  Self-reported items on the baseline survey. Some of these demographic variables will also be considered covariates in analyses.
Demographic moderators: education | 3 months
  Self-reported items on the baseline survey. Some of these demographic variables will also be considered covariates in analyses.
Demographic moderators: marital status | 3 months
  Self-reported items on the baseline survey. Some of these demographic variables will also be considered covariates in analyses.
Demographic moderators: retirement status | 3 months
  Self-reported items on the baseline survey. Some of these demographic variables will also be considered covariates in analyses.

OTHER OUTCOMES:
Mitochondrial functioning biomarkers | 3 months
  Targeted metabolomic measurement of ~300 plasma metabolites (e.g., amino acids, acylcarnitines, organic acids), primarily associated with mitochondrial biochemical pathways
Epigenetic DNA modification profile | 3 months
  Measurement of DNA methylation in peripheral blood monocytes (PBMCs) to determine "bio-age" and Apparent Methylomic Aging Rate (AMAR)
Epigenetic microRNA biomarkers | 3 months
  Measurement of microRNA populations in blood (PBMCs and endothelial cell microparticles) using Hi-Seq
Vascular environment/endothelial functioning biomarker 1 | 3 months
  Measurement of plasma biomarkers of systemic inflammation (C-reactive protein (CRP))
Vascular environment/endothelial functioning biomarker 2 | 3 months
  Measurement of endothelial cell adhesiveness and activation (vascular adhesion molecule 1 (sVCAM-1))
Vascular environment/endothelial functioning biomarker 3 | 3 months
  Measurement of endothelial cell adhesiveness and activation (intercellular adhesion molecule 1 (sICAM-1))
Vascular environment/endothelial functioning biomarker 4 | 3 months
  Measurement of endothelial cell adhesiveness and activation (P- and E-selectins)
Vascular environment/endothelial functioning biomarker 5 | 3 months
  Measurement of oxidative stress (F2-isoprostane)
Vascular environment/endothelial functioning biomarker 6 | 3 months
  Measurement of coagulation (fibrinogen)
Glucoregulatory and lipid metabolism biomarker 1 | 3 months
  Measurement of fasting plasma insulin
Glucoregulatory and lipid metabolism biomarker 2 | 3 months
  Measurement of glucose
Glucoregulatory and lipid metabolism biomarker 3 | 3 months
  Measurement of lipid panel components (total cholesterol, LDL, HDL and triglycerides)
Glucoregulatory and lipid metabolism biomarker 4 | 3 months
  Measurement of hemoglobin A1c (HbA1c)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Allison, MDD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - South Bay Latino Research Center, Chula Vista, California
  - UCSD, San Diego, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with universities or centers in AHA funded research networks.

REFERENCES:
- [Background] Andresen EM, Malmgren JA, Carter WB, Patrick DL. Screening for depression in well older adults: evaluation of a short form of the CES-D (Center for Epidemiologic Studies Depression Scale). Am J Prev Med. 1994 Mar-Apr;10(2):77-84. PMID 8037935
- [Background] Gardiner PA. Understanding and influencing sedentary behaviour in older adults [dissertation]. Vol Doctorate of Philosophy. Brisbane, Australia: University of Queeensland; 2011.
- [Background] Salmon J, Hume C, Ball K, Booth M, Crawford D. Individual, social and home environment determinants of change in children's television viewing: the Switch-Play intervention. J Sci Med Sport. 2006 Oct;9(5):378-87. doi: 10.1016/j.jsams.2006.06.018. Epub 2006 Aug 14. PMID 16908215
- [Background] Norman GJ, Sallis JF, Gaskins R. Comparability and reliability of paper- and computer-based measures of psychosocial constructs for adolescent physical activity and sedentary behaviors. Res Q Exerc Sport. 2005 Sep;76(3):315-23. doi: 10.1080/02701367.2005.10599302. PMID 16270708
- [Background] Norman G, Vaughn AA, Roesch S, Sallis JF, Calfas K, Patrick K. Development of decisional balance and self-efficacy measures for adolescent sedentary behaviors. Psychology and Health 2004;19:561-575.
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Rosenberg DE, Sallis JF, Kerr J, Maher J, Norman GJ, Durant N, Harris SK, Saelens BE. Brief scales to assess physical activity and sedentary equipment in the home. Int J Behav Nutr Phys Act. 2010 Jan 31;7:10. doi: 10.1186/1479-5868-7-10. PMID 20181057
- [Derived] Takemoto M, Schechtman M, Villa N, Talavera G, Sears DD, Natarajan L, Owen N, Rosenberg DE, Dunstan D, Allison M, Kerr J. Arriba por la Vida Estudio (AVE): Study protocol for a standing intervention targeting postmenopausal Latinas. Contemp Clin Trials. 2019 Apr;79:66-72. doi: 10.1016/j.cct.2019.02.004. Epub 2019 Feb 13. PMID 30771560